CLINICAL TRIAL: NCT05487118
Title: Effects of Photobiomodulation Therapy (LASER) Associated With Motor Control Exercises for Chronic Non-specific Low Back Pain
Brief Title: PBMT Associated With MCE for Chronic Non- Specific Low Back Pain
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Collaborators: University of Bergen (Other)
Responsible Party: Principal Investigator, Ernesto Cesar Pinto Leal Junior, Full professor, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 5.289.714
Record Dates: First submitted 2022-08-02; First posted 2022-08-04 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Low Back Pain
Keywords: Photobiomodulation Therapy; LLLT; Motor Control Exercise
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo PBMT + MCE (Placebo Comparator): Placebo photobiomodulation therapy (PBMT), with a dose of 0 J, will be applied before a protocol of motor control exercises (MCE).
  Interventions: Device: Placebo PBMT + MCE
- Active PBMT + MCE (Active Comparator): Active photobiomodulation therapy (PBMT), with a dose of 30 J, will be applied before a protocol of motor control exercises (MCE).
  Interventions: Device: Active PBMT + MCE

INTERVENTIONS:
Device: Placebo PBMT + MCE — Placebo PBMT will be irradiated at 4 sites in the lumbar region and 6 sites in the patient's abdominal region, without any emission of therapeutic dose. After, the patient will be submitted to a MCE protocol consisting on stabilization exercises and isometric abdominal training. The treatment will be performed twice a week (on non-consecutive days), for 6 weeks, yielding 12 treatment sessions.
  Arms: Placebo PBMT + MCE
Device: Active PBMT + MCE — Active PBMT will be irradiated at 4 sites in the lumbar region and 6 sites in the patient's abdominal region, with a dose of 30 J per site. After, the patient will be submitted to a MCE protocol consisting on stabilization exercises and isometric abdominal training. The treatment will be performed twice a week (on non-consecutive days), for 6 weeks, yielding 12 treatment sessions.
  Arms: Active PBMT + MCE

SUMMARY:
Non-specific low back pain (LBP) is a very prevalent health condition and is highly associated with disability worldwide. There is evidence that patients with non-specific LBP may have impairments in the control of postural muscles. In this way, motor control exercises (MCE) may be an interesting alternative in the treatment of patients with non-specific LBP. In addition, the association of MCE and photobiomodulation therapy (PBMT) may potentiate its benefits, since PBMT has ergogenic effects. Therefore, the aim of this study is to evaluate the ergogenic effects of PBMT, using low-level laser therapy, when associated with MCE in patients with chronic non-specific low back pain.

DETAILED DESCRIPTION:
This is a randomized, triple-blind (patients, therapists, outcome assessors), placebo-controlled trial, with voluntary patients with chronic non-specific low back pain. One hundred and forty-eight patients will be randomly allocated to two treatment groups: Placebo PBMT associated with MCE or Active PBMT associated with MCE. Treatment will be performed twice a week (on non-consecutive days), for 6 weeks, yielding 12 treatment sessions. Placebo PBMT or Active PBMT will be applied before the MCE protocol.

The clinical outcomes will be obtained at the end of treatment (6 weeks), one month after the end of treatment, 3, 6 and 12 months after randomization. The biochemical outcome will be obtained only after the end of treatment. The remaining outcomes will be obtained after the end of treatment, one month after the end of treatment, 3, 6 and 12 months after randomization.

The data will be collected by a blinded assessor. The statistical analysis will follow the intention-to-treat principles and the between-group differences will be calculated using two-way repeated measures ANOVA.

The project was also approved by the Research Ethics Committee from Universidade Nove de Julho, under the number 5.289.714.

Board Affiliation: Comissão Nacional de Ética em Pesquisa (CONEP) Phone: +55113385-9010 - Email: comitedeetica@uninove.br Address: Vergueiro nº 235/249. Liberdade, Sao Paulo, Sao Paulo, Brazil

ELIGIBILITY:
Inclusion Criteria:

* patients seeking care for chronic non-specific low back pain (defined as pain or discomfort between the costal margins and the inferior gluteal folds, with or without referred symptoms in the lower limbs, for at least 3 month);
* with a pain intensity of at least 3 points measured by a 0-10 points pain numerical rating scale;
* aged between 18 and 65 years;
* able to read Portuguese.

Exclusion Criteria:

* evidence of nerve root compromise (i.e. one or more of motor, reflex or sensation deficit);
* serious spinal pathology (such as fracture, tumor, inflammatory and infectious diseases);
* patients with severe skin diseases (eg, skin cancer, erysipelas, severe eczema, severe dermatitis, severe psoriasis and severe hives lupus);
* decompensated severe cardiovascular and metabolic diseases;
* previous back surgery;
* patients with cancer;
* body mass index (BMI) ≥ 30.
* pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2022-08-22 (Actual); Primary Completion 2024-03-04 (Actual); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | At the end of treatment (6 weeks after randomization)
  Pain intensity will be measured by Pain Numerical Rating Scale that evaluates pain intensity levels perceived by the patient on an 11-point scale ranging from 0 to 10, with 0 being 'no pain' and 10 'the worst possible pain'. Higher scores mean worse outcome.
Disability | At the end of treatment (6 weeks after randomization)
  Disability will be measured by the 24-item Roland Morris Disability Questionnaire. The questionnaire consists of 24 items that patient has to answer 'yes' or 'no'. The minimum value is 0 and the maximum value is 24. Higher scores mean worse outcome.

SECONDARY OUTCOMES:
Pain intensity | 1 month after the end of the treatment, 3, 6 and 12 months after randomization
  Pain intensity will be measured by Pain Numerical Rating Scale that evaluates pain intensity levels perceived by the patient on an 11-point scale ranging from 0 to 10, with 0 being 'no pain' and 10 'the worst possible pain'. Higher scores mean worse outcome.
Disability | 1 month after the end of the treatment, 3, 6 and 12 months after randomization
  Disability will be measured by the 24-item Roland Morris Disability Questionnaire. The questionnaire consists of 24 items that patient has to answer 'yes' or 'no'. The minimum value is 0 and the maximum value is 24. Higher scores mean worse outcome.
Levels of prostaglandin E2 (PGE2) | At the end of treatment (6 weeks after randomization)
  Levels of PGE2 will be measured by blood samples
Medication intake | At the end of treatment (6 weeks after randomization), 1 month after the end of treatment, 3, 6 and 12 months after randomization
  The medication intake will be measured from self-report
Co-interventions | At the end of treatment (6 weeks after randomization),1 month after the end of treatment, 3, 6 and 12 months after randomization
  Co-interventions will be measured from self-report
Adverse events | At the end of treatment (6 weeks after randomization), 1 month after the end of treatment, 3, 6 and 12 months after randomization
  Adverse events will be measured from self-report

CONTACTS AND LOCATIONS:
Overall Officials: Shaiane Tomazoni, PhD, Principal Investigator — University of Bergen
Locations (2):
- Brazil (2):
  - Santa Casa de Misericórdia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Laboratory of Phototherapy and Innovative Technologies in Health, São Paulo

IPD SHARING:
Plan to Share IPD: Yes
The IPD will be available on reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will become available during five years after the study completion
Access Criteria: All IPD that underlie results in a publication will be available on reasonable request.

REFERENCES:
- [Derived] de Oliveira MFD, Bjordal JM, Schardong J, Plentz RDM, Casalechi HL, Leal-Junior ECP, Tomazoni SS. Effects of photobiomodulation therapy associated with motor control exercise for chronic non-specific low back pain: protocol for a randomised placebo-controlled trial. BMJ Open Sport Exerc Med. 2024 Sep 26;10(3):e002199. doi: 10.1136/bmjsem-2024-002199. eCollection 2024. PMID 39345834